CLINICAL TRIAL: NCT03202992
Title: Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of Topical ABI-1968 in Subjects With Anal High-Grade Squamous Intraepithelial Lesions (aHSIL)
Brief Title: Study of Topical ABI-1968 in Subjects With Precancerous Anal Lesions Resulting From Human Papillomavirus (HPV) Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antiva Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABI-1968-201
Record Dates: First submitted 2017-06-24; First posted 2017-06-29 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: HSIL, High-Grade Squamous Intraepithelial Lesions; Human Papilloma Virus Infection; HIV Infection; Anal Cancer; Anus Neoplasms
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Papillomavirus Infections; HIV Infections; Anus Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 2 Phases: Part A, up to 5 cohorts of 3 subjects each will receive a single dose of ABI-1968 Topical Cream. In Part B, three cohorts (3 subjects per cohort) will receive multiple doses in 3 ascending dose strengths of ABI-1968 Topical Cream. After completing the ascending dose multiple-dosing cohorts, a multiple-dosing Cohort Expansion group of 30 subjects will be initiated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Dose 1 -Single Ascending Dose (SAD) (Experimental): SAD Dose Level 1 of ABI-1968 topical cream applied on Day 1 of the study
  Interventions: Drug: ABI-1968
- Dose 2 -Single Ascending Dose (SAD) (Experimental): SAD Dose Level 2 of ABI-1968 topical cream applied on Day 1 of the study
  Interventions: Drug: ABI-1968
- Dose 3 -Single Ascending Dose(SAD) (Experimental): SAD Dose Level 3 of ABI-1968 topical cream applied on Day 1 of the study
  Interventions: Drug: ABI-1968
- Dose 4 -Single Ascending Dose(SAD) (Experimental): SAD Dose Level 4 of ABI-1968 topical cream applied on Day 1 of the study
  Interventions: Drug: ABI-1968
- Dose 5 -Single Ascending Dose(SAD) (Experimental): SAD Dose Level 5 of ABI-1968 topical cream applied on Day 1 of the study
  Interventions: Drug: ABI-1968
- Dose 1 - Multiple Ascending Dose(MAD) (Experimental): MAD Dose Level 1 of ABI-1968 topical cream applied at Day 1, Day 8, Day 15, Day 22 and Day 29
  Interventions: Drug: ABI-1968
- Dose 2 -Multiple Ascending Dose(MAD) (Experimental): MAD Dose Level 2 of ABI-1968 topical cream applied at Day 1, Day 8, Day 15, Day 22 and Day 29
  Interventions: Drug: ABI-1968
- Dose 3 -Multiple Ascending Dose(MAD) (Experimental): MAD Dose Level 3 of ABI-1968 topical cream applied at Day 1, Day 8, Day 15, Day 22 and Day 29
  Interventions: Drug: ABI-1968
- Multiple Ascending Dose (MAD) Cohort Expansion (Experimental): MAD Cohort Expansion of ABI-1968 applied at Day 1, Day 8, Day 15, Day 22 and Day 29
  Interventions: Drug: ABI-1968
- Dose 4-Multiple Ascending Dose(MAD) (Experimental): MAD Dose Level 3 of ABI-1968 topical cream applied at Day 1, Day 8, Day 15, Day 22 and Day 29
  Interventions: Drug: ABI-1968

INTERVENTIONS:
Drug: ABI-1968 — Topical cream applied at Day 1 for the SAD portion and applied at Day 1, Day 8, Day 15, Day 22 and Day 29 for the MAD portion

SUMMARY:
This study evaluates the use of ABI-1968, a topical cream, in the treatment of anal precancerous lesions in adults with and without human immunodeficiency virus (HIV) infection.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects, at least 27 years old.
2. Confirmed diagnosis of intra-anal HSIL at least 3 months prior to screening and confirmed by histopathology (with p16 positive staining)
3. Intra-anal HSIL are visible and evaluable by HRA at the time of screening, and no lesion(s) is suspicious for invasive cancer.
4. For HIV-positive subjects, CD4 count must be at least 200/mm3 with undetectable (<50 copies/mL) viral load within the 3 months prior to enrollment. Subjects must be on a stable regimen of antiretroviral drugs for the 3 months prior to enrollment.

Exclusion Criteria:

1. Women who are pregnant, plan to become pregnant in the next 3 months, or lactating females.
2. Received topical treatment or ablative procedures for aHSIL in the 6 months prior to enrolment.
3. History of cancer, including anal cancer (with the exception of basal cell or squamous cell carcinoma of the skin), or currently undergoing treatment for any skin cancer.
4. History of genital herpes with > 3 outbreaks per year.
5. Plan to have excision or ablation of the lesion(s) within 3 months of enrolment.

Min Age: 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ABI-1968 for the treatment of aHSIL | SAD portion is 29 days/MAD portion is 84 days
  Number of participants with Adverse Events related to treatment

SECONDARY OUTCOMES:
Systemic exposure to ABI-1968 Topical Cream following topical application to the anal canal. | SAD portion is 29 days/MAD portion is 84 days
  Plasma concentrations of ABI-1968 over time
Histopathology of areas with biopsy-proven disease following single and multiple doses of ABI-1968 Topical Cream. | SAD portion is 29 days/MAD portion is 84 days
  Number of subjects with complete and or partial regression of aHSIL by High Resolution Anoscopy (HRA) and histopathology

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Chair — Choosing to participate in a study is an important personal decision. Talk with your doctor and family members or friends about deciding to join a study. To learn more about this study, you or your doctor may use the contacts provided below.
Locations (6):
- United States (5):
  - Research Center, San Francisco, California
  - Research Center, Orlando, Florida
  - Research Center, Chicago, Illinois
  - Research Center, New York, New York
  - Research Center, Winston-Salem, North Carolina
- Research Center, Sydney, Darlinghurst, Australia

IPD SHARING:
Plan to Share IPD: No